CLINICAL TRIAL: NCT02977325
Title: Translation and Cultural Adaptation of the Arthritis Self-Efficacy Scale
Brief Title: Validation of the Questionnaire ASES
Acronym: ASES
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Clermont Communauté (Other); Innovatherm (Industry)
Responsible Party: Sponsor
Other Study IDs: CHU-0293
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Knee Osteoarthritis; Physical Activity; Education; Self-management; Exercise
Keywords: Physical activity level; Personal efficacy; Knee osteoarthritis; Self-management; Self-care; Education and exercise in knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Physical activity: One group participated in therapeutic programs centered on the physical activity
  Interventions: Other: water cure
- water cure exclusively: This group followed exclusively the water cure
  Interventions: Other: water cure

INTERVENTIONS:
Other: water cure

SUMMARY:
Questionnaires are often irreplaceable tools of collection of information in research and in the clinical practice. Coupled with other measures, they can be simple complementary tools, but questionnaires are sometimes the only way to collect data, such as self-service efficacy.

The objective of this study is a validation of the French translation of the ASES. To guarantee the comparability between the original version and the translated version, the translation of a questionnaire supposes two essential stages: a literal translation and an adaptation to the cultural context, to the habits of life and to the idioms of the target population. This new version will afterward be validated with patient's troop.

DETAILED DESCRIPTION:
The investigators are particularly interested in the Arthritis Self-Efficacy Scale (ASES), conceived to highlight a change of the faith of the patients in their capacities to make usual thinks or behaviour in front of consequences of the degenerative osteoarthritis, further to a therapeutic education.

The ASES is an auto-questionnaire compound of 20 items, from 0 to 10 on a digital scale and distributed in three domains: control of the pain (on 50), function (on 90) and other symptoms (on 60).

This questionnaire was already translated into Swedish, Dutch and Turkish.

Translation of the ASES and cultural adaptation :

The translation of the ASES in French followed the recommendations of the literature, which recommend a double translation, then a double back - translation with synthesis of the data in every stage. A final commission deliberate then a final translation, culturally adapted.

Patients' cohort and procedure of validation :

The prospective validation will be made with patients affected by degenerative osteoarthritis who fill the questionnaire ASES. These patients arose from cures of three thermal establishments of Auvergne. One group participated in therapeutic programs centered on the physical activity; the other one followed exclusively the water cure and received at the end of the cure an explanatory notebook on the degenerative osteoarthritis with physical exercises centered on the muscular strengthening of lower limbs.

Feedback :

Assessments conducted by the using of self - questionnaires:

- Sent by mail to the patients and back at 3 and 3,5 months

Ethics:

A written consent was collected before inclusion in the study and a document intended for the information was given to the patient. The study is anonymous, indeed, index forms will be coded before IT processing to guarantee the anonymity of the patient.

ELIGIBILITY:
Inclusion criteria :

Both sexes, 50-75 years old Knee osteoarthritis Patients affiliated to a social security scheme Patients realizing a Spa Therapy Acceptance to participate in the study

Exclusion criteria :

< 50-year-old patients or > 75 years Inflammatory, tumoral, traumatic or infectious rheumatism Cardiac decompensation Disorders of the concentration or the compression of the written or oral French language.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with knee osteoarthritis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-07; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
personal efficacy by means of the French questionnaire ASES "Arthritis Self-Efficacy Scale" | at 3 months
personal efficacy by means of the French questionnaire ASES "Arthritis Self-Efficacy Scale" | at 3 months +15 days

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel COUDEYRE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France